CLINICAL TRIAL: NCT05308225
Title: A Phase 1b/2a, Open-Label, Dose-Escalation Study of the Safety and Efficacy of an Anti-CD38 Antibody Drug Conjugate (STI-6129) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Study to Assess Anti-CD38 Antibody Drug Conjugate in Relapsed or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 38ADC-RRMM-101
Record Dates: First submitted 2022-03-15; First posted 2022-04-04 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; relapsed refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: To determine DLT and MTD, the design uses a 3+3 design for the dose-escalation stage.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STI-6129 (Experimental): Seven dosing cohorts will be evaluated: 0.67 mg/kg, 0.88 mg/kg, 1.18 mg/kg, 1.56 mg/kg, 2.08 mg/kg, 2.77 mg/kg, 3.68 mg/kg where STI-6129 will be intravenously administered once as part of a 4-week treatment cycle.
  Interventions: Biological: STI-6129

INTERVENTIONS:
Biological: STI-6129 — Anti-CD38 A2 human antibody drug conjugate (ADC) containing an antibody covalently bound to a duostatin tubulin inhibitor

SUMMARY:
This is a two-stage phase 1b/2a, open-label, multicenter, dose-escalation study of STI-6129 administered intravenously once in a 4-week cycle in subjects with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a two-stage phase 1b/2a, open-label, multicenter, dose-escalation study of STI-6129 administered intravenously once in a 4-week cycle in subjects with relapsed or refractory multiple myeloma.

The study is designed to identify the recommended phase 2 dose (RP2D) of STI-6129 by assessing the safety, preliminary efficacy and pharmacokinetics using a conventional 3+3 study design for dose escalation in stage one and then the second stage will be an expansion study to assess preliminary efficacy.

Patients will be enrolled sequentially within each cohort and between cohorts during the dose escalation portion of the study with a 28-day cycle of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have relapsed or refractory multiple myeloma (RRMM) after having received prior lines of anti-myeloma treatments, including being refractory to a proteasome inhibitor, immunomodulatory agent and an anti-CD38 monoclonal antibody
* Measurable disease as defined by one of the following: abnormal serum or M-protein levels; abnormal serum free light chain (FLC) assay; ≥ 30% clonal plasma cells in the bone marrow aspirate or biopsy sample
* Pulse oximetry ≥ 92% on room air
* Eastern Cooperative Oncology Group (ECOG) performance of 0 - 2
* Be willing and able to comply with the study schedule and all study requirements
* Willing to follow contraception guidelines

Exclusion Criteria:

* Prior systemic anti-tumor therapy or an investigational drug within 5 half-lives or 4 weeks of D1, whichever is shorter, preceding the first dose of study drug
* Prior treatment with allogeneic hematopoietic stem cell transplantation within 6 months, has active graft versus host disease following transplant or currently receiving immunosuppressive therapy following transplant
* Diagnosis of other malignancies if the malignancy required therapy in the last 3 years or is not in complete remission
* Current history of CTCAE Grade 3 muscle paresis or ocular disorders that are Grade 3 or 2
* Has any clinically significant low baseline lab results for hemoglobin, platelet counts, and neutrophil counts at screening
* Abnormal INR or aPTT, unless on a stable dose of an anticoagulant
* Has ≥ Grade 3 neuropathy or Grade 2 neuropathy with associated pain
* Has any clinically significant baseline lab results for creatinine clearance, serum aspartate aminotransferase, alanine aminotransferase, total bilirubin
* New York Heart Association Class > 2
* Left ventricular ejection fraction < 40%
* Prolonged QTcF interval on a 12-lead electrocardiogram
* Has active COVID-19 infection, and not present with symptoms within 4 weeks of study drug
* Has an active bacterial, viral, or fungal infection
* Has known HIV or acquired immunodeficiency syndrome-related illness, acute or history of chronic hepatitis B or C
* Is currently pregnant or breast feeding or planning on either during the study
* Has any significant medical condition, abnormality, or psychiatric illness that would prevent study participation
* Has any additional clinical history that would place the patient at an unacceptable risk if the patient participates in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Safety of STI-6129 | Baseline through study completion at up to approximately 24 months
  Safety as assessed by incidence of adverse events (AEs), severe AEs (SAEs), DLTs, neurotoxicity and laboratory abnormalities using the Common Terminology Criteria for Adverse Events (CTCAE Version 5)

SECONDARY OUTCOMES:
Measuring Pharmacokinetic [PK] Profile | Baseline through study completion at up to approximately 24 months
  STI-6129 blood plasma concentrations will be measured for the total antibody plus conjugated toxin (STI 6129) and the free toxin
Overall response and duration | Baseline through study completion at up to approximately 24 months
  Response and duration determined according to the International Myeloma Working Group (IMWG) response criteria
Assess preliminary efficacy | Baseline through study completion at up to approximately 24 months
  As a measure of activity, overall response rate will be assessed according to the modified International Myeloma Working Group (IMWG) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Rajshekar Chakraborty, MD, Principal Investigator — Columbia University; David Kaminetzky, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - NYU Lagone Health, New York, New York
  - Columbia University Medical Center, New York, New York
  - Gabrail Cancer Center, Canton, Ohio